Official Title: A web-based intuitive eating intervention for young women with disordered eating: A pilot randomized controlled trial

**NCT number:** not yet assigned

**Date of document: 2/15/2021** 

## Informed Consent

Jayne Duncan, M. A. and Dr. Charles Swencionis, Ph.D. of Yeshiva University (YU) in Bronx, New York, along with a team of graduate students are conducting a study investigating the impact of a 10-week online intervention focused on intuitive eating on health outcomes, and psychological flexibility. If you are a woman between the ages of 18 and 30, reside in the United States or Canada, and do not currently meet the criteria for an eating disorder we invite you to participate in this study. The screening questionnaires you completed put you in a "high risk" category, meaning that you are more likely to have negative body image and problems with food, and therefore you are invited to participate.

If you opt to participate, you will be randomly assigned to either undergo a 10-week online intervention or to a wait-list group. If you are in the intervention group, you will participate by reading short articles, watching videos, and engaging in question-and-answer sessions once per week for 10 consecutive weeks. You will answer a series of questionnaires at the beginning and end of the 10-week intervention so its efficacy can be tested. If you are in the wait-list group you will complete a series of questionnaires at the beginning and end of a 10-week interval, so we can compare changes in those who completed the intervention versus those who did not. You will be invited to participate in the intervention after your time on the wait-list.

All of your personal data (i.e. survey responses, weight/height, anything typed/sent as a part of the intervention) will be ANONYMOUS. We will use randomly generated numerical identifiers to protect your identity and confidentiality. The code "name" you provide is required on this form only in order to prevent duplicate participation; your responses will NOT be linked with your identity. This study is the subject of a thesis project in the Summer of 2020, and potentially will also be the subject of a journal publication/s. Under no circumstances will your personal information ever be a focus of attention or will your name or identifying characteristics appear in writing in connection with this project. The research team will secure and ultimately dispose of the information.

Please indicate below that you have read this form and whether or not you consent to participation. The study has been approved by Western IRB. If you have any further questions about the study, please contact study investegator Jayne Duncan, M. A. at jduncan1@mail.yu.edu or study supervisor Dr. Charles Swencionis at charles.swencionis@yu.edu . If you have concerns about the study, you can contact the chair of Western IRB at help@wirb.com or (800) 562-4789.

Sincerely, Jayne Duncan, M. A. Dr. Charles Swencionis, Ph.D.

-----

After reading the above, I hereby voluntarily consent to participate in this study. I am aware that I have the right to withdraw from this study at any time without penalty.